CLINICAL TRIAL: NCT06022718
Title: A Randomised Crossover Comparison of Kinesio-Taping and Rigid-Taping on Vertical Jump in Individuals With Pes Planus
Brief Title: Comparison of Kinesio-Taping and Rigid-Taping on Vertical Jump in Individuals With Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EKK21-22/016/006
Record Dates: First submitted 2023-08-26; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Pes Planus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: Low dye bandage technique was used with a 3.8 cm wide rigid band (Leuko® Sportstape Premium, Germany) for rigid taping. RT was performed on both feet in the subtalar neutral position while participants in the prone position with their heels and feet out of the bed. The taping protocol described elsewhere was followed. To optimise rigid tape adhesion, feet were washed and dried before taping. To increase consistency, the same researcher (MU) applied all taping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio-taping Group (Experimental): Kinesio® Tex GoldFP (USA) was applied on both feet in the prone position with the knee extended, and the feet in a slightly plantar flexed position and hanging off the bed. The first Kinesio-taping was cut as an I shape and prepared for the transverse arch ligament correction technique. The non-stretched starting anchor was attached to the dorsum of the 5th metatars on the lateral side of the foot, passed from the plantar surface to the medial side with 75-100% tension. The non-stretched end was attached to the medial side of the ankle over the navicular region. The non-stretched initial anchor of the second Kinesio-taping strip starting from the proximal dorsal of the 5th. metatarsal on the lateral side of the foot.
  Interventions: Other: Taping
- Rigid-taping Group (Experimental): Low dye bandage technique was used with a 3.8 cm wide rigid band (Leuko® Sportstape Premium, Germany) for rigid taping. Rigid taping was performed on both feet in the subtalar neutral position while participants in the prone position with their heels and feet out of the bed. The taping protocol described elsewhere was followed. 21 To optimise rigid tape adhesion, feet were washed and dried before taping. To increase consistency, the same researcher (MU) applied all taping.
  Interventions: Other: Taping

INTERVENTIONS:
Other: Taping — Kinesio taping and Rigid taping was applied.

SUMMARY:
The effects of Kinesio-taping and rigid-taping on vertical jump performance have been investigated; however, results remain unclear.

DETAILED DESCRIPTION:
The effect of Kinesio-taping and rigid-taping on controlling foot pronation remains unclear due to contradicted results. Moreover, to our knowledge, there is not any study to elucidate the effect of rigid-taping on vertical jump performance. Therefore, the investigators hypothesised that rigid-taping would be more effective on vertical jump performance because of its direct mechanical correction in pes planus, and the study was aimed to compare the effects of Kinesio-taping and RT on vertical jump performance in sedentary adults with pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals between the ages of 18-35,
* Individuals without any chronic disease

Exclusion Criteria:

* Those with lower extremity injuries in the last 1 year,
* Those with a history of lower extremity surgery and visual or vestibular disorders,
* Those with other foot deformities accompanying pes planus,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Vertical Jump | 2 minutes
  The jumping performance of each participant was evaluated using the VertiMetric (Lafayette Instrument Company, Lafayette, IN) device.
Foot Posture | 10 minutes
  Foot Posture Index is used for clinical diagnostic purposes that evaluate whether a foot is in pronation, supination, or normal posture. The sum of six-item scores between 0-5 are interpreted as normal foot, scores of 6-12 as pes planus, and scores <0 as pes cavus.

SECONDARY OUTCOMES:
Physical Activity | 3 minutes
  The physical activity levels of the participants were evaluated with the International Physical Activity Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Salih Angın, PhD., Study Chair — Cyprus International University
Locations (1):
- Mehmet Miçooğulları, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledoux WR, Hillstrom HJ. The distributed plantar vertical force of neutrally aligned and pes planus feet. Gait Posture. 2002 Feb;15(1):1-9. doi: 10.1016/s0966-6362(01)00165-5. PMID 11809575
- [Background] Razeghi M, Batt ME. Foot type classification: a critical review of current methods. Gait Posture. 2002 Jun;15(3):282-91. doi: 10.1016/s0966-6362(01)00151-5. PMID 11983503
- [Background] Aguilar MB, Abian-Vicen J, Halstead J, Gijon-Nogueron G. Effectiveness of neuromuscular taping on pronated foot posture and walking plantar pressures in amateur runners. J Sci Med Sport. 2016 Apr;19(4):348-53. doi: 10.1016/j.jsams.2015.04.004. Epub 2015 Apr 24. PMID 25956688
- [Background] Arastoo AA, Aghdam EM, Habibi AH, Zahednejad S. Kinetic factors of vertical jumping for heading a ball in flexible flatfooted amateur soccer players with and without insole adoption. Prosthet Orthot Int. 2014 Jun;38(3):204-10. doi: 10.1177/0309364613492790. Epub 2013 Jul 4. PMID 23828877
- [Background] Vanezis A, Lees A. A biomechanical analysis of good and poor performers of the vertical jump. Ergonomics. 2005 Sep 15-Nov 15;48(11-14):1594-603. doi: 10.1080/00140130500101262. PMID 16338725
- [Background] Nakajima MA, Baldridge C. The effect of kinesio(R) tape on vertical jump and dynamic postural control. Int J Sports Phys Ther. 2013 Aug;8(4):393-406. PMID 24175126
- [Background] Franettovich MM, Murley GS, David BS, Bird AR. A comparison of augmented low-Dye taping and ankle bracing on lower limb muscle activity during walking in adults with flat-arched foot posture. J Sci Med Sport. 2012 Jan;15(1):8-13. doi: 10.1016/j.jsams.2011.05.009. Epub 2011 Aug 30. PMID 21880545
- [Background] Angin S, Crofts G, Mickle KJ, Nester CJ. Ultrasound evaluation of foot muscles and plantar fascia in pes planus. Gait Posture. 2014;40(1):48-52. doi: 10.1016/j.gaitpost.2014.02.008. Epub 2014 Feb 26. PMID 24630465